CLINICAL TRIAL: NCT04620304
Title: A Phase I, Open-Label, Multi-Dose Study for Evaluation of the Safety, Pharmacokinetics, and Antiviral Activity of UB-421 Subcutaneous Formulation Administered in HIV-1 Infected Treatment Naive Patients
Brief Title: Study for Evaluation of the Safety, Pharmacokinetics, and Antiviral Activity of UB-421 Subcutaneous Formulation Administered in HIV-1 Infected Treatment Naive Patients
Status: Completed | Phase: Phase 1 | Type: Interventional
Sponsor: United BioPharma (Industry)
Collaborators: Kaohsiung Medical University Chung-Ho Memorial Hospital (Other); Kaohsiung Veterans General Hospital. (Other); Taoyuan General Hospital (Other Government)
Responsible Party: Sponsor
Allocation: Non-Randomized | Model: Sequential | Masking: None | Purpose: Treatment
Other Study IDs: UBP-A122-HIV
Record Dates: First submitted 2020-10-22; First posted 2020-11-06 (Actual); Last update posted 2023-04-24 (Actual); Status verified 2023-04

CONDITIONS: HIV-1 Infection

STUDY DESIGN:
Oversight: Data Monitoring Committee: Yes | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (3):
- Cohort A (Experimental): receive 4 weekly fixed doses of UB-421 SC at 250 mg
  Interventions: Biological: UB-421 SC(dB4C7C22-6 mAb)
- Cohort B (Experimental): receive 4 weekly fixed doses of UB-421 SC at 500 mg
  Interventions: Biological: UB-421 SC(dB4C7C22-6 mAb)
- Cohort C (Experimental): receive 4 weekly fixed doses of UB-421 SC at 700 mg
  Interventions: Biological: UB-421 SC(dB4C7C22-6 mAb)

INTERVENTIONS:
Biological: UB-421 SC(dB4C7C22-6 mAb) — The UB-421 SC (dB4C7C22-6 mAb) will be supplied at a concentration of 125 mg/mL after reconstitution. Subjects will receive weekly UB-421 SC injections during the 4-week Treatment Period.

SUMMARY:
This is a phase I, open-label, dose-escalation study to investigate short-term safety, pharmacokinetics, and antiviral activity of UB-421 SC with 4 weekly doses in treatment naive HIV-1 infected patients. Eligible (n=6 per dose cohort) subjects will be sequentially enrolled into 3 escalating-dose cohorts to receive 4 weekly fixed doses of UB-421 SC at either 250 mg (Cohort A), 500 mg (Cohort B) or 700 mg (Cohort C). Subjects should be followed for safety for additional 4 weeks after the last UB-421 SC dosing. In order to control viral load while minimizing confounding in safety assessment, subjects can initiate standard anti-retroviral therapy (ART) two weeks after the last UB-421 SC dosing.

Escalation to the next higher dose cohort will be determined based on dose limited toxicity (DLT) evaluation. The dose escalation will be stopped if ≥ 2/6 subjects experience DLT or when clinical trial steering committee (CTSC) determines it is not suitable to escalate the dose level.

In this study, DLT is defined as any ≥ grade 3 AE occurred within 21 days from prior UB-421 SC dosing and is considered drug related.

When there is any ≥grade 3 AE(s) occurred within 21 days from prior UB-421 SC dosing in any subject out of the current dose cohort (n=6), the duty of the CTSC will be initiated. The CTSC will be responsible for DLT evaluation. The committee members will evaluate the safety data of all subjects in each cohort through baseline to at least 21 days following the last UB-421 SC dosing. The administration of the next higher dose level at TV1 will be conducted after the committee grants the dose escalation. However, dose escalation will be proceeded if there is no ≥ grade 3 AE and upon agreement from all investigators without holding the steering committee meeting.

Subjects will be assessed at Screening, weekly during Treatment Period and Follow-up Period. The assessment includes physical examination, vital sign, laboratory parameters, HIV-1 viral load, CD4+ and CD8+ T-cell counts. Samples for the drug concentration measurement will be collected at weekly intervals throughout the study, immediately before UB-421 SC dosing. Additional intensive PK sampling will be scheduled during the first dosing interval (from TV1 to TV2) at 1, 3, 6, 24, 48, 72 and 96 hours post first UB-421 SC dosing for PK subgroup (at least 3 subjects per dose cohort). The immunogenicity of UB-421 SC will be monitored by measuring anti-UB-421 antibodies in pre-dose serum samples at day 0 and post-dose serum at day 14, 28, 35, 42 and 49. Viral reservoir, immunophenotyping and CD4+ (D1) receptor occupancy will also be explored.

Subjects should discontinue from UB-421 SC treatment if they experience a sustained decrease from baseline in CD4+ (D2) T cell counts of ≧50% at two consecutive visits or drug-related AE(s) with severity grade 3 or 4 (according to the Division of AIDS, National Institute of Allergy and Infectious Diseases (DAIDS) AE grading).

ELIGIBILITY:
Inclusion Criteria:

1. HIV-1 seropositive, with documented HIV-1 infection by official, signed, written history (e.g. laboratory report);
2. Male and female, age 20 years or older;
3. Asymptomatic (generalized lymphadenopathy can be included), defined as subjects without stage 3 defining opportunistic illnesses according to revised Surveillance Case Definition for HIV Infection published in 2014, which was determined by the Investigator based on the medical history, physical examination, ECG, and laboratory evaluations;
4. CD4+ (D1) T cell count > 350 cells/mm3 at the Screening Visit;
5. HIV-1 viral load > 5,000 copies/mL at the Screening Visit;
6. HIV antiretroviral therapy (ART)-naïve i.e., subjects who receive no prior or current HIV antiretroviral drugs;
7. Male subjects and female subjects of childbearing potential must agree to use the acceptable method of contraception during the course of the study (excluding women who are not of childbearing potential). Women of childbearing potential (WOCBP) must have a negative serum pregnancy test at the Screening Visit; Definitions Women NOT of childbearing potential: women who are permanently or surgically sterilized or postmenopausal. Permanent sterilization includes hysterectomy, and/or bilateral oophorectomy, and/or bilateral salpingectomy and/or tubal ligation.

   Postmenopausal women: 12 months of amenorrhea in a woman over age 45 years in the absence of other biological or physiological causes.

   Acceptable method of birth control for WOCBP: abstinence; implant; intrauterine device; hormonal contraceptive (injectable, oral contraceptives, transdermal patches, or contraceptive rings) plus barrier method (male condom, female condom or diaphragm).

   Acceptable method of birth control for male subjects: abstinence; condom.
8. Subjects signed the informed consent before undergoing any study procedures. -

Exclusion Criteria:

1. Females who are pregnant, lactating, or breastfeeding, or who plan to become pregnant during the study;
2. Subjects with acute opportunistic infection(s) or bacterial infection(s), that the delayed initiation of ART would not be allowed, as judged by the Investigator;
3. Any stage 3 defining opportunistic illnesses such as Kaposi's sarcoma according to the revised Surveillance Case Definition for HIV Infection published in 2014 within the past 12 months before the Screening Visit;
4. Serious illness requiring systemic treatment and/or hospitalization for at least 7 days prior to the Screening Visit;
5. Any previous exposure to a monoclonal antibody within 12 weeks prior to the Screening Visit;
6. Any previous hypersensitivity reaction to monoclonal antibody;
7. Any significant diseases (other than HIV-1 infection) or clinically significant findings that, in the Investigator's judgment, would potentially compromise study compliance or the ability to evaluate safety/efficacy;
8. Current or chronic history of liver disease, or known hepatic or biliary abnormalities (with the exception of Gilbert's syndrome or asymptomatic gallstones);
9. Presence of hepatitis B surface antigen (HBsAg) or positive hepatitis C antibody test within 12 weeks prior to the Screening Visit;
10. Serum GPT/ALT value is 3 times or greater than the upper limit of normal (≥ 3 xULN) at the Screening Visit;
11. Serum GOT/AST value is 3 times or greater than the upper limit of normal (≥ 3 xULN) at the Screening Visit;
12. Serum total bilirubin (TBIL) value is 1.5 times or greater than the upper limit of normal (≥1.5 xULN) at the Screening Visit;
13. Serum creatinine value is greater than 1.3 times the upper limit of normal (>1.3xULN) at the Screening Visit;
14. Any vaccination within 8 weeks prior to the Screening Visit;
15. Any treatment with immunomodulators, such as interleukins, interferon, cyclosporine, systemic corticosteroid, or systemic chemotherapy within 12 weeks prior to the Screening Visit; Note: Subjects received short-term low dose oral (i.e. prednisone ≤0.5mg/kg/day for ≤ 1-month duration), inhaled, nasal, or topical steroids will not be excluded.
16. Prior participation in any HIV vaccine trial;
17. Subjects who have ever received UB-421 IV or SC formulations;
18. Receipt of other investigational study agent within 12 weeks before the Screening Visit;
19. Life expectancy of less than 12 months;
20. Any current alcohol or illicit drug use that, in the Investigator's opinion, would interfere with the subject's ability to comply with the dosing and visit schedules and protocol evaluations.

    -

Min Age: 20 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 15 (Actual)
Dates: Start 2021-01-01 (Actual); Primary Completion 2022-05-25 (Actual); Study Completion 2022-05-25 (Actual)

PRIMARY OUTCOMES:
Numbers and incidence of TEAEs | 28 days
  Numbers and incidence of TEAEs that are ≥ Grade 2 and study treatment related, TEAEs (any grades) by maximum severity, TEAEs by relationship to study treatment, SAEs, TEAEs leading to death, and TEAEs leading to discontinuation of study treatment will be tabulated by dose cohort and will be summarized by system organ class and preferred term for study period (Treatment or Follow-up). The "Division of AIDS (DAIDS) Table for Grading the Severity of Adult and Pediatric Adverse Events" will be used in this study for all AE severity grading, except skin abnormalities, which will be evaluated according to Common Terminology Criteria for Adverse Events (CTCAE).

SECONDARY OUTCOMES:
The virologic responses during the Treatment Period | 28 days
  The proportion of subjects ever achieving HIV-1 RNA reduction > X log10 copies/mL;
Pharmacokinetics (PK) of UB-421 SC | 28 days
  • Ctrough for each dosing interval
Pharmacokinetics (PK) of UB-421 SC | 28 days
  Cmax of first dosing interval;
Pharmacokinetics (PK) of UB-421 SC | 28 days
  AUC0-inf (if applicable).
The virologic responses during the Treatment Period (from TV1 to EOT) | 28 days
  The proportion of subjects with virologic rebound

OTHER OUTCOMES:
Serum anti UB-421 antibody leve | 49 days
  Serum levels of anti-UB-421 antibody

CONTACTS AND LOCATIONS:
Locations (1):
- Kaohsiung Veterans General Hospital, Kaohsiung City, Taiwan